CLINICAL TRIAL: NCT04199949
Title: Effects of Five Days of Physical Inactivity on Endothelial Function in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Moira Taylor, Dr Moira A Taylor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: A90355
Record Dates: First submitted 2019-11-19; First posted 2019-12-16 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: FMD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 5 consecutive days of normal daily levels of physical activity and matched food intake
- Inactivity (Experimental): 5 consecutive days of reduced step count by 80% compared to the Control trial, whilst placing the non-dominant arm in a sling, and reduced food intake (~ 20%) to match the reduction in energy expenditure induced by inactivity
  Interventions: Behavioral: Inactivity

INTERVENTIONS:
Behavioral: Inactivity — On days 1 and 6 of each main trial, the participants will be asked to attend the laboratory after an overnight fast of at least 8 to 12h to undergo brachial and popliteal arteries FMD measurements (30 min apart) using duplex-Doppler ultrasound, followed by assessment of the hand grip strength of their non-dominant hand using a hand dynamometer.
  Arms: Inactivity

SUMMARY:
Physical inactivity is a significant predictor of major non-communicable diseases such as type 2 diabetes (7%), cardiovascular disease (6%), musculoskeletal disorders and some types of cancer, and has been proposed to be the 4th leading cause of death worldwide. The investigators aim is to assess the vascular (endothelial) function before and after a 5-day period of reduced activity of upper and lower limbs via an arm sling and daily step counts reduction, respectively, in healthy participants. Twelve young (ages of 18 - 35 years), healthy, males and females, recreationally active with a body mass index between 18 and 27 kg/m2 will be recruited. The participants will then randomly undergo two 5-day interventions: (A) 5 consecutive days of habitual daily levels of physical activity and matched food intake (Control trial). (B) 5 consecutive days of reduced step count by 80% compared to the Control trial combined with their non-dominant arm placed in a sling and a reduction in food (energy) intake (~20%) to match the reduction in energy expenditure induced by inactivity (Inactivity trial). On days 1 and 6 of each experimental trial, the endothelial function of the brachial and popliteal arteries, and hand grip strength will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Males
* Age (18-35 years old)
* Body mass index (BMI) of 18-27 kg/m2
* Recreationally active
* Ability to give informed consent

Exclusion Criteria:

* Smoking
* Any metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism) or cardiovascular (e.g. heart or blood) abnormalities including hypertension or heart failure
* Clinically significant abnormalities on screening including ECG abnormalities
* Taking routine medication that may alter cardiovascular function and blood flow (e.g. blood pressure-lowering drugs or drugs that cause hypertension)
* Well-trained individuals
* On an energy-restricted diet or seeking to lose weight
* High alcohol consumption (<3-4 units/day)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of flow-mediated vasodilatation (FMD) of the brachial artery | Over 6 minutes and 20 seconds on day 1 and day 6 of each study arm
  The FMD of the brachial artery will be measured using an ultrasound collected at baseline and continuously for 80 seconds post-arm occlusion for 5 minutes
Change from baseline of flow-mediated vasodilatation (FMD) of the popliteal artery | Over 6 minutes and 20 seconds on day 1 and day 6 of each study arm
  The FMD of the popliteal artery will be measured using an ultrasound collected at baseline and continuously for 80 seconds post-arm occlusion for 5 minutes

SECONDARY OUTCOMES:
Hand grip strength | 3 minutes
  The hand grip strength will be measured using a hand dynamometer. Three maximum hand grips separated by one minute rest at the end of each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No